CLINICAL TRIAL: NCT05676814
Title: Pecto-intercostal Fascial Block With Perineural Adjuvants for Postoperative Analgesia Following Sternotomy in Patients Undergoing Cardiac Surgery
Brief Title: Pecto-intercostal Fascial Block (PIFB) for Postop Analgesia Following Sternotomy in Cardiac Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00090669
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-04

CONDITIONS: Analgesia; Sternotomy
Keywords: Pecto-intercostal Fascial Block; Postoperative; Pain; Cardiac Surgery
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be blinded to their treatment arm assignment, as will all research personnel who be responsible for collection of outcome data, as well as the surgeons performing the procedure, and critical care staff caring for the patients in the postoperative period. The anesthesiologist who will be performing the Pecto-intercostal Fascial Block (PIFB) will open the envelope informing them of the arm assignment; they will be the only care providers unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pecto-intercostal Fascial Block (PIFB) (Active Comparator): Subjects in this arm receive standard of care PIFB after surgery
  Interventions: Drug: Pecto-intercostal Fascial Block (PIFB)
- PIFB with adjuvants (Experimental): Subjects in this arm receive standard of care PIFB with additional medications after surgery
  Interventions: Drug: PIFB with adjuvants

INTERVENTIONS:
Drug: Pecto-intercostal Fascial Block (PIFB) — PIFB done with bupivacaine and epinephrine
  Arms: Pecto-intercostal Fascial Block (PIFB)
Drug: PIFB with adjuvants — PIFB with bupivacaine, epinephrine, clonidine, and dexamethasone
  Arms: PIFB with adjuvants

SUMMARY:
The purpose of this randomized, triple-blinded, prospective, feasibility study is to compare postoperative analgesia provided by Pecto-intercostal Fascial Block (PIFB) when performed with local anesthetic solution with or without perineural adjuvants in patients following cardiac surgery involving sternotomy. The study team hypothesizes that the patients receiving PIFB with bupivacaine with epinephrine, clonidine, and dexamethasone will have lower dynamic pain over the first 36 hours compared to those receiving PIFB with just bupivacaine and epinephrine.

DETAILED DESCRIPTION:
This will be a randomized, triple-blinded, prospective, feasibility trial. Written informed consent will be obtained from all study participants prior to randomization. Patients scheduled to undergo cardiac surgery involving sternotomy at Atrium Health Wake Forest Baptist will be screened for eligibility. These patients will be approached for enrollment by research staff either during their preoperative assessment clinic visit prior to their surgery date, or when admitted as inpatients and scheduled for surgery. Subjects chosen to participate will be randomized into one or other arm and PIFB will be performed after skin closure and before transport from the operating room to the ICU. For patients who are randomized at enrollment but later excluded due to exclusion criteria prior to block placement, their randomization assignment will be replaced at the end of the initial recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Adults between undergoing cardiac surgery involving sternotomy

Exclusion Criteria:

* Patients with any contraindications to regional anesthesia, such as history of allergy to amide local anesthetics or any of the perineural adjuvants
* existing neurologic deficit in the chest wall;
* remaining intubated at the six hour point after block placement
* weight under 50kg
* undergoing emergency surgical procedures or urgent return to the operating room
* active endocarditis or mediastinitis
* moderate to severe right ventricular function before or after cardiopulmonary bypass
* reliance on mechanical circulatory support devices, such as intra-aortic balloon pump or Impella
* reliance on extracorporeal membrane oxygenation
* localized or systemic infection
* chronic use of high dose opioid analgesics (defined as daily use greater than 30 oral morphine milligram equivalents (OMME) for over one month prior to surgery)
* those who are pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Coleman, DO, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Started | 16 | 15
Completed | 12 | 8
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 12 | 8 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) Pain Score - Based on Patient-reported Dynamic Numerical Rating Scale (NRS) Pain Scores
Description: Based on patient-reported dynamic Numerical Rating Scale (NRS) pain scores with incentive spirometer (IS) use in subjects that are extubated. Pain scores range from 0 to 10 with higher scores denoting more pain. 0 to 6 hrs after placement.
Time Frame: 0 to 6 hours after block placement
Measure: Mean (Standard Deviation); unit: scores on a scale*hour
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 12 | 8
scores on a scale*hour | 6.39 (3.23) | 4.22 (3.76)

2. Primary Outcome: Area Under the Curve (AUC) Pain Score - Based on Patient-reported Dynamic Numerical Rating Scale (NRS) Pain Scores
Description: Based on patient-reported dynamic NRS pain scores with incentive spirometer (IS) use in subjects that are extubated. Pain scores range from 0 to 10 with higher scores denoting more pain.
Time Frame: 12 hours after block placement
Measure: Mean (Standard Deviation); unit: scores on a scale*hour
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 12 | 8
scores on a scale*hour | 3.28 (2.03) | 4.06 (3.65)

3. Primary Outcome: Area Under the Curve (AUC) Pain Score - Based on Patient-reported Dynamic Numerical Rating Scale (NRS) Pain Scores
Description: as for outcome 2
Time Frame: 18 hours after block placement
Measure: Mean (Standard Deviation); unit: scores on a scale*hour
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 12 | 8
scores on a scale*hour | 4.00 (2.09) | 5.12 (3.23)

4. Primary Outcome: Area Under the Curve (AUC) Pain Score - Based on Patient-reported Dynamic Numerical Rating Scale (NRS) Pain Scores
Description: as for outcome 2
Time Frame: 24 hours after block placement
Measure: Mean (Standard Deviation); unit: scores on a scale*hour
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 12 | 8
scores on a scale*hour | 3.18 (2.19) | 4.71 (3.06)

5. Primary Outcome: Area Under the Curve (AUC) Pain Score - Based on Patient-reported Dynamic Numerical Rating Scale (NRS) Pain Scores
Description: as for outcome 2
Time Frame: 36 hours after block placement
Population: data wasn't collected
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Patient-reported Numerical Rating Scale (NRS) Pain Scores at Rest
Description: Pain scores range from 0 to 10 with higher scores denoting more pain.
Time Frame: 6 hours after block placement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 12 | 8
units on a scale | 5.25 (3.22) | 3.43 (4.24)

7. Secondary Outcome: Patient-reported Numerical Rating Scale (NRS) Pain Scores at Rest
Description: Pain scores range from 0 to 10 with higher scores denoting more pain.
Time Frame: 6, 12, 18, 24 hours after block placement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 12 | 8
units on a scale
  6 hour | 5.25 (3.22) | 3.43 (4.24)
  12 hour | 2.67 (2.02) | 3.14 (3.18)
  18 hour | 2.45 (2.42) | 3.5 (3.25)
  24 hour | 3.09 (2.26) | 3.5 (3.78)

8. Secondary Outcome: Average Cumulative Opioid Consumption
Description: Average Cumulative Opioid Consumption in milligrams
Time Frame: 36 hours after block placement
Population: data wasn't collected
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Average Time to First Opioid Administration
Description: Average Time to First Opioid Administration - Postoperative after extubation measured in minutes
Time Frame: Up to 36 hours after block placement
Population: data not collected
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Average Time to Extubation
Description: Average Time to Extubation - measured in minutes
Time Frame: Up to 36 hours after block placement
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 12 | 8
Minutes | 276.815 (78.609) | 232.020 (68.689)

11. Secondary Outcome: Duration of Intensive Care Unit (ICU) Admission
Description: Duration of Intensive Care Unit (ICU) Admission - measured in Average number of hours.
Time Frame: Up to 52 hours after block placement
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 12 | 8
Hours | 50.620 (32.302) | 51.541 (59.249)

12. Secondary Outcome: Incentive Spirometry Volumes
Description: An incentive spirometer is a handheld medical device that measures the volume of subject's breath. The volume of air displaced is indicated in milliliters on a scale located on the device enclosure. This device measures what is called vital capacity, the amount of air that is breathed in and out of the lungs.
Time Frame: 6, 12, 18, 24 hours after block placement
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 12 | 8
Milliliters
  Baseline | 2750 (823.43) | 3427.08 (743.27)
  6 hours | 525 (338.56) | 1333.33 (857.97)
  12 hours | 968.06 (287.14) | 1519.44 (716.12)
  18 hours | 878.79 (336.08) | 1440.63 (794.07)
  24 hours | 1093.94 (337.25) | 1275 (498.65)

13. Secondary Outcome: Safety Outcome: Nausea Incidence
Description: Average number of incidences of Nausea
Time Frame: Up to 36 hours after block placement
Population: data wasn't collected
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Safety Outcome: Vomiting Incidence
Description: Average number of Vomiting incidences
Time Frame: Up to 36 hours after block placement
Population: data wasn't collected
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Safety Outcome: Postoperative Delirium Incidence
Description: Average number of Delirium incidences
Time Frame: Up to 36 hours after block placement
Population: data wasn't collected
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Numeric Rating Scale (NRS) Satisfaction With the Analgesic Regimen
Description: Patient-reported scores range from 0-10 where 0 represents completely unsatisfied and 10 represents completely satisfied.
Time Frame: 36 hours after block placement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
Number analyzed (Participants) | 12 | 8
units on a scale | 7.92 (1.98) | 8.88 (.99)

ADVERSE EVENTS:
Time Frame: up to 36 hours postop
Arm/Group | Pecto-intercostal Fascial Block (PIFB) | PIFB With Adjuvants
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT05676814/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT05676814/ICF_000.pdf